CLINICAL TRIAL: NCT01901796
Title: Integrated Maternal Psychosocial Assessment to Care Trial (IMPACT): Intervening Early to Improve Maternal and Family Well-being.
Brief Title: Integrated Maternal Psychosocial Assessment to Care Trial (IMPACT) Full Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Norlien Foundation (Other); Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Principal Investigator, Dawn Kingston, Associate Professor, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 00036912
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; CBT
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening and CBT (Experimental): Screening and Cognitive Behavioral Therapy. The intervention group will be screened and if they need criteria they will complete the 6, 30-minute online, interactive CBT modules over 6 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Usual care (No Intervention): Usual prenatal care

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy- an effective, non-pharmacological treatment for depression and anxiety.
  Arms: Screening and CBT

SUMMARY:
We hypothesize that the intervention will: (1) offer a feasible approach for providing mental healthcare to pregnant women and have a high level of acceptability by pregnant women and healthcare providers; (2) reduce symptoms of depression, stress, anxiety, and parenting stress; improve parenting competence, coping, and relationship adjustment compared to usual care; and (3) reduce the risk of poor maternal-infant attachment. As such, this early intervention holds promise for reducing maternal mental health morbidity and its negative influences on infants, children, and families.

DETAILED DESCRIPTION:
One of the main reasons that women do not receive treatment is that their mood and anxiety problems are not detected. Despite recommendations and high rates of acceptance by providers and women, only a minority of providers conduct psychosocial assessments as part of routine prenatal care. Computer-based 'screening' is an acceptable and feasible approach to assessment of sensitive issues including prenatal and postnatal intimate partner violence, mental health problems, and postpartum depression by patients and providers. It is well-suited for busy clinical settings and is advantageous in that it offers a consistent approach to assessment, is resource-sparing, can be tailored to meet the specific needs of patients, can be used with audio/video for low literacy, provides a real-time summary for patients/providers,achieves similar or higher rates of disclosure of violence and mental health problems, and is preferred by patients because they perceive it as more anonymous compared to interviews or questionnaires.

However, psychosocial assessment on its own is ineffective in preventing or treating mood disorders and unethical in the absence of treatment options. As such, many providers do not assess pregnant women for mood disorders because non-pharmacological treatments are frequently unavailable and pregnant women prefer them. Cognitive behavioural therapy (CBT) is a highly effective, non-pharmacological treatment for depression and anxiety and is recommended by perinatal national Australian guidelines as a potentially effective EARLY intervention for reducing the risk of maternal-child outcomes.

ELIGIBILITY:
Inclusion criteria:

Pregnant women will be eligible for Phase 2 if they are:

1. < 28 weeks gestation (to provide the opportunity to complete 6 modules and follow-up questionnaires prior to delivery)
2. able to speak/read English; and (3) willing to complete email questionnaires

Exclusion Criteria:

1. >28 weeks gestation
2. unable to speak/read English
3. unable to complete email questionnaires

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study is the feasibility/acceptability of integrated psychosocial care and its components. | 6 weeks post randomization
  Feasibility/acceptability of the intervention will be assessed through individual face-to-face or telephone-based semi-structured qualitative interviews of both clinic staff and women in the intervention group. The field does not allow for all questions to be provided. Sample question for clinic staff is 'What aspects made it easy/challenging to use the tablet for prenatal assessment as part of routine prenatal care?' Sample questions for intervention group participants: 1)How did you feel about answering these kinds of questions on a tablet?; 2)Please describe any concerns you had about answering these questions on a tablet; 3)How would you prefer the results to be shared with you

SECONDARY OUTCOMES:
Maternal depression, anxiety, stress | on recruitment, 6 weeks post randomization and 3 months postpartum
  Depression, Anxiety, and Stress Scale (DASS-21) Self-reported by mother on emailed questionnaire
Maternal coping | on recruitment, 6 weeks post-randomization and 3 months postpartum
  The Brief Cope Self-reported by mother on emailed questionnaire
Relationship Adjustment | on recruitment, 6 weeks post-randomization and 3 months postpartum
  Scale: Dyadic Adjustment Scale, DAS-7 Self-reported by mother on emailed questionnaire
Parenting Stress | 3 months postpartum
  Parenting Stress Scale Self-reported by mother
Parenting competence | 3 months postpartum
  Parenting Sense of Competence Scale Self-reported by mother on emailed questionnaire
Maternal-infant attachment | 3 months postpartum
  Maternal Attachment Inventory (MAI) Self-reported by mother on emailed questionnaire
Trait anxiety | on recruitment, 6 weeks postrandomization, 3 months postpartum
  State Trait Anxiety Inventory (STAI) Self-reported by mother on emailed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dawn A Kingston, Ph.D, Principal Investigator — University of Calgary
Locations (1):
- Westview Health Centre, Stony Plain, Alberta, Canada

REFERENCES:
- [Derived] Bright KS, Stuart S, Mcneil DA, Murray L, Kingston DE. Feasibility and Acceptability of Internet-Based Interpersonal Psychotherapy for Stress, Anxiety, and Depression in Prenatal Women: Thematic Analysis. JMIR Form Res. 2022 Jun 10;6(6):e23879. doi: 10.2196/23879. PMID 35687403
- [Derived] Bright KS, Mughal MK, Wajid A, Lane-Smith M, Murray L, Roy N, Van Zanten SV, Mcneil DA, Stuart S, Kingston D. Internet-based interpersonal psychotherapy for stress, anxiety, and depression in prenatal women: study protocol for a pilot randomized controlled trial. Trials. 2019 Dec 30;20(1):814. doi: 10.1186/s13063-019-3897-z. PMID 31888712
- [Derived] Kingston D, Austin MP, Hegadoren K, McDonald S, Lasiuk G, McDonald S, Heaman M, Biringer A, Sword W, Giallo R, Patel T, Lane-Smith M, van Zanten SV. Study protocol for a randomized, controlled, superiority trial comparing the clinical and cost- effectiveness of integrated online mental health assessment-referral-care in pregnancy to usual prenatal care on prenatal and postnatal mental health and infant health and development: the Integrated Maternal Psychosocial Assessment to Care Trial (IMPACT). Trials. 2014 Mar 6;15:72. doi: 10.1186/1745-6215-15-72. PMID 24597683